CLINICAL TRIAL: NCT01075828
Title: A Korean Post Marketing Surveillance Study On Erbitux® (Cetuximab) In Patients With Locally Advanced or Recurrent and/or Metastatic Squamous Cell Cancer of the Head and Neck (SCCHN)
Brief Title: Prospective, Post Marketing Surveillance Study On Erbitux® (Cetuximab) in Patients With Locally Advanced or Recurrent and/or Metastatic Squamous Cell Cancer of the Head and Neck in Korea
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Other Study IDs: EMR62241-508 (EMR 62202-551)
Record Dates: First submitted 2010-02-24; First posted 2010-02-25 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-08

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck Neoplasms; Neoplasms, Squamous Cell; Cetuximab
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasms, Squamous Cell | interventions — Cetuximab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Cetuximab — Subjects will be treated according to the national label of cetuximab in combination with radiation therapy.
  Other Names: Erbitux

SUMMARY:
After consultation with the Korean Health Authorities, the two Post-Authorization Safety Studies EMR 62202-509 (NCT01082315) and EMR 62241-508 (NCT01075828) were combined within one study protocol EMR 062202-551. This Post-Marketing Surveillance Study (PMS) EMR 062202-551 is requested by the Korean Health Authorities to continue monitoring of Erbitux and provide further information about safety and toxicity in clinical practice in at least 900 patients during 6 years.

All data points from the EMR 62202-509 (NCT01082315) and EMR 62241-508 (NCT01075828) remain unchanged in protocol EMR 062202-551. Therefore, the Sponsor has decided not to separately disclose the EMR 062202-551 study titled "A Korean Post-Marketing Surveillance Study On Erbitux® (Cetuximab) in Patients With Locally Advanced or Recurrent and/or Metastatic Squamous Cell Cancer of the Head and Neck (originally EMR 62241-508) and in Patients With EGFR-expressing, KRAS wild-type Metastatic Colorectal Cancer (originally EMR 62202-509)" on clinicaltrials.gov.

DETAILED DESCRIPTION:
This is a prospective, Post Marketing Surveillance (PMS) study on Erbitux® (Cetuximab) in patients with locally advanced or recurrent and/or metastatic squamous cell cancer of the head and neck in Korea

This prospective study will collect safety information from more than 300 subjects treated with Erbitux as final evaluable cases. During the PMS period, subject background, subject's medical (surgery, anti-cancer treatment) history, Erbitux treatment status, concurrent medication, response evaluation, status and reason of discontinuation, all adverse events (AEs; regardless of the causal relationship to Erbitux), and abnormal results of laboratory tests will be collected for the study purpose.

The PMS is based on all cases treated with Erbitux at least once. The PMS will be done within 6 years from the approval date of the new indication. This PMS is requested by the Korean Regulatory Authorities. After approval of new indication in Korea, it is further required to investigate more than 300 subjects during 6 years according to local regulations to continue monitoring and provide further information about safety and toxicity in clinical practice.

OBJECTIVES Analysis on safety and efficacy information on the use of Erbitux in the market and factors affecting its safety and efficacy.

Primary objective:

* To obtain safety information on the use of Erbitux in subjects with locally advanced SCCHN or recurrent and/or metastatic in terms of frequency and severity of AEs

Secondary objectives:

* To gather clinical efficacy information of the treatment

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are eligible for Erbitux treatment according to the indication in the national label of Erbitux. The national label approved by Korea Food & Drug Administration is "Erbitux in combination with radiation therapy is indicated for the treatment of subjects with locally advanced or recurrent and/or metastatic SCCHN

Exclusion Criteria:

* Subjects who are not eligible for Erbitux treatment according to the indication in the national label of Erbitux

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with locally advanced or recurrent and/or metastatic SCCHN eligible for Erbitux treatment will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 221 (Actual)
Dates: Start 2009-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Frequency of Adverse Events | 6 years
  The frequency and severity of all adverse events, regardless of the causal relationship to Erbitux, will be measured within 6 years of the observational period from the approval date of the new indication

SECONDARY OUTCOMES:
Clinical efficacy | 6 years
  The duration of control of locoregional disease, 1-year/2-year/3-year locoregional control rate, best tumor response will be measured within the observational period from the approval date of the new indication

CONTACTS AND LOCATIONS:
Locations (1):
- Chungnam National University Hospital, Jung-gu Daejeon, South Korea